CLINICAL TRIAL: NCT00006143
Title: A Randomized, Open-Label Study of Recombinant Human Growth Hormone (r-hGH) in Children With HIV-Associated Growth Failure
Brief Title: Growth Hormone Treatment of Children With HIV-Associated Growth Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: P1011; 11646 (Registry Identifier: DAIDS ES); ACTG P1011; PACTG P1011
Record Dates: First submitted 2000-08-07; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Outcome; serostim; Developmental Disabilities
MeSH Terms: conditions — HIV Infections; Developmental Disabilities | interventions — Human Growth Hormone

INTERVENTIONS:
Drug: Somatropin

SUMMARY:
The purpose of this study is to determine the effectiveness of recombinant human growth hormone (r-hGH) on growth in HIV-infected children.

Studies have shown that HIV-infected children do not grow at a normal rate and are shorter than HIV-uninfected children who are the same age. Growth hormone has been used for many years to treat children with growth hormone deficiency and has been safe and effective in helping them to grow normally. The growth hormone to be used in this study, r-hGH, is an investigational hormone (not yet approved by the Food and Drug Administration [FDA]) made in the laboratory. It has helped HIV-positive adults gain weight and improve their physical performance. This study has been changed to include a needle-free device for drug delivery which will improve patient comfort and acceptability. Patients will no longer receive growth hormone through traditional needles but through a needle-free device.

DETAILED DESCRIPTION:
Wasting, or loss of lean tissue, is a serious consequence of AIDS. Body composition findings in HIV-infected children are similar to those of HIV-uninfected children with classic growth hormone deficiency. Evidence suggests that therapeutic administration of growth hormone (GH) can induce anabolic effects, reverse pathologic catabolism, and perhaps even improve immune function. As survival to adolescence and beyond improves with modern therapy in children with HIV infection, it will become increasingly important to address the problems of stunting and short stature in this population. [AS PER AMENDMENT 09/04/01: Recent evidence suggests that needle-free delivery is preferred by young children below the age of ten years. Given the advantages of a needle-free delivery system for the administration of growth hormone, most significantly the reduction of risk for HIV contaminated needle-stick injuries to care providers and other household members, it has been decided to use this method of study drug delivery for all study participants.]

Children are assigned randomly to 1 of the following treatment groups:

Group 1: Children receive a single dose of r-hGH once a day. Group 2: Children receive half the dose of r-hGH that Group 1 receives, once a day.

Group 3a: Children receive no r-hGH for the first 24 weeks [AS PER AMENDMENT 01/03/01: 48 weeks] of the study. After Week 24 [AS PER AMENDMENT 01/03/01: Week 48], they receive the same dose as that of Group 1.

Group 3b: Children receive no r-hGH for the first 24 weeks [AS PER AMENDMENT 01/03/01: 48 weeks] of the study. After Week 24 [AS PER AMENDMENT 01/03/01: Week 48], they receive the same dose as that of Group 2.

Subcutaneous injections are administered [AS PER AMENDMENT 09/04/01: using a needle-free device], daily for 96 weeks in Groups 1 and 2; after 24 weeks [AS PER AMENDMENT 01/03/01: 48 weeks] on study, the treatment-delayed control group (Group 3) receives injections for 72 weeks [AS PER AMENDMENT 01/03/01: 48 weeks]. The first injection is at the clinic and parents/guardians are trained how to prepare and administer the injections. Children are closely monitored for toxicity, with dosing adjustments if needed. Evaluations and laboratory tests are done at clinic visits every 4 weeks to determine growth indicators, body chemistries, CD4 cell counts, HIV-1 RNA PCR, and anti-hGH antibodies and for routine hematology testing, dietary intake assessment, and MRI scans. [AS PER AMENDMENT 01/03/01: MRI scans are no longer performed.]

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are 4 to 12 years of age for girls, and 4 to 13 years of age for boys (consent of parent/guardian is required).
* Are HIV-positive.
* Are not growing normally.
* Have a normal intake of food each day.
* Are able to walk.
* Have been on stable anti-HIV therapy for at least 24 weeks before study entry and will continue therapy for the entire duration of the study with no anticipated change in therapy for the first 48 weeks of the study. (These therapy requirements reflect a change.)
* Are willing and able to follow study requirements.

Exclusion Criteria

Children may not be eligible for this study if they:

* Had steady fever of 101 degrees F or higher during the 2 weeks before study entry.
* Have a serious infection requiring medications within 30 days prior to study entry.
* Are being fed through a vein.
* Have severe diarrhea, intestinal bleeding or blockage, or are unable to absorb food.
* Have cancer.
* Have taken medications that may interfere with the study drug or have had radiation.
* Have diabetes or a history of sugar intolerance.
* Have carpal tunnel syndrome (unless it has been surgically repaired).
* Have heart or kidney problems, or serious swelling of any kind.
* Have any condition other than HIV infections that may have affected growth or that makes it difficult to measure height.
* Have any known allergies to the study drug.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102
Dates: Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harland Winter, Study Chair; Wayne Dankner, Study Chair
Locations (20):
- United States (18):
  - Phoenix Children's Hosp., Phoenix, Arizona
  - Childrens Hosp. LA - Dept. of Ped., Div. of Clinical Immunology & Allergy, Los Angeles, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - South Florida CDC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Chicago Children's CRS, Chicago, Illinois
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr., The Bronx, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Texas Children's Hosp. CRS, Houston, Texas
  - VCU Health Systems, Dept. of Peds, Richmond, Virginia
- Puerto Rico (2):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan